CLINICAL TRIAL: NCT01737372
Title: A Pilot Study to Assess microRNA Biomarkers in Early and Later Stage Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: John F. Foley, MD (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, John F. Foley, MD, President and Sponsor-Investigator, Rocky Mountain MS Research Group, LLC
Organization: Rocky Mountain MS Research Group, LLC (Other)
Other Study IDs: 003-001-GEN
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Clinically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid and blood may be stored for future immunological, cell product and microRNA testing related to the primary outcome of the this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Secondary Progressive MS (SPMS): Secondary Progressive MS participants
- Clinically Isolated Syndrome (CIS): Clinically isolated syndrome participants
- Healthy participants: No immunological or neurological illnesses.

SUMMARY:
This study will look at the blood and cerebrospinal fluid of consented participants who either have early stage multiple sclerosis (clinically isolated syndrome) or who have later stage (secondary progressive multiple sclerosis), or participants who do not have any neurological or autoimmune illness. Biomarkers and microRNA will be assessed for group differences.

DETAILED DESCRIPTION:
Multiple Sclerosis is a chronic autoimmune disorder of the central nervous system. While there are current immunomodulatory therapies that have been shown to be efficacious in the early stages of MS, these therapies are less potent in the later phases of MS. We can look at magnetic resonance imaging with gadolinium to measure active disease but it does not detect axonal degeneration. Therefore, there is a need to identify other biomarkers that may be used to diagnose MS and predict disease progression. Biomarkers found in the cerebrospinal fluid (CSF) are in closer proximity to the inflammatory lesion sites and are more sensitive.

This pilot study seeks to characterize differences in microRNA profiles and cell products in the early and later stages of MS, with the hope that that microRNA profiles could then be correlated to clinical and CSF inflammation indexes. CSF will be obtained from 45 participants.

ELIGIBILITY:
Inclusion Criteria:

* able to understand and agree to informed consent;
* male or female patients 18-68 years of age
* no disease modifying therapy 60 days prior to Baseline
* EDSS score of less than or equal to 3.0 if a CIS patient; or less than or equal to 7.5 if SPMS patient
* Labs within normal range no greater than 2 times the ULN or at the discretion of the PI
* weight 46 kilograms to 127 kilograms inclusive
* no active systemic infection
* not currently pregnant or breast feeding
* no history of corticosteroid treatment or relapse within 60 days prior to Baseline.

Exclusion Criteria:

* not able to understand informed consent
* if any of the inclusion criteria is not met
* HIV infection, or current active Hepatitis B or C infection, positive HCVAb or HBsAG or HBcAB
* positive pregnancy test
* patient withdraws consent
* Coumadin use within 60 days prior to Baseline

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 45 participants will be enrolled into a study to examine the microRNA and cell products profile in both cerebrospinal fluid (CSF) and blood. Study population will consist of a total of: 20 CIS patients defined as patients having a single attack (or the appearance of one or more symptoms characteristic of MS) high risk of developing MS, when no other diseases or causes are apparent.
  20 SPMS patients 5 normal, non-diseased controls
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To characterize differences in microRNA profile and cell product patterns between early and later stage multiple sclerosis. | baseline

SECONDARY OUTCOMES:
Correlate microRNA profiles with clinical and CSF inflammation indexes | baseline

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — Rocky Mountain MS Research Group, LLC
Locations (1):
- Rocky Mountain MS Clinic, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No